CLINICAL TRIAL: NCT05403554
Title: A Phase 1, Open-Label, Dose Finding Study of NI-1801, a Bispecific Mesothelin X CD47 Engaging Antibody, As a Single Agent, in Combination with Anti-PD-1 Antibody, and in Combination with Weekly Paclitaxel (Standard of Care) in Patients with Mesothelin Expressing Ovarian, Pancreatic, Non-Small-Cell-Lung and Triple-Negative Breast Cancers
Brief Title: A Study of NI-1801 in Patients with Mesothelin Expressing Solid Cancers
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Light Chain Bioscience - Novimmune SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCB-1801-001; 2021-003808-40 (EudraCT Number)
Record Dates: First submitted 2022-05-24; First posted 2022-06-03 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-09

CONDITIONS: Epithelial Ovarian Cancer; Triple Negative Breast Cancer; Non-squamous Non-small-cell Lung Cancer; Pancreatic Adenocarcinoma (ductal Adenocarcinoma); Endometrioid Ovarian Cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Triple Negative Breast Neoplasms | interventions — pembrolizumab; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- NI-1801 Single Agent (Experimental): NI-1801 will be evaluated in patients with MSLN-expressing advanced, metastatic solid tumors
  Interventions: Drug: Biological NI-1801
- NI-1801 in Combination with Pembrolizumab (Experimental): NI-1801 will be evaluated in patients with MSLN-expressing advanced, metastatic solid tumors in combination with anti-PD-1 antibody
  Interventions: Drug: NI-1801 in combination with anti-PD1 (Pembrolizumab)
- Randomized cohort (Active Comparator): In the randomized, open-label cohort design, the experimental arm will receive the investigational drug NI-1801 at the P2RD in combination with weekly administration of paclitaxel (80 mg/m^2) over 4-week cycles.
  Interventions: Drug: NI-1801 in combination with paclitaxel; Drug: Paclitaxel

INTERVENTIONS:
Drug: Biological NI-1801 — Treatment will be administered in 28-day cycles for up to 12 months until disease progression, unacceptable toxicity, or Investigator/patient decision to withdraw study consent. Each subject will receive the assigned dose of NI-1801 on Cycle 1, Day 1. Subsequent doses will be given Q2W, which may be adjusted to every three weeks if recommended from the ongoing PK/PD model analysis.
  Arms: NI-1801 Single Agent
Drug: NI-1801 in combination with anti-PD1 (Pembrolizumab) — In the combination with pembrolizumab cohort, the starting NI-1801 dose will be 300 mg. Pembrolizumab will be administered at the dosage of 400 mg every 6 weeks, in 4 cycles. Pembrolizumab will be administered as first drug; later, NI-1801 will be infused after 30 minutes.
  Arms: NI-1801 in Combination with Pembrolizumab
Drug: NI-1801 in combination with paclitaxel — The experimental arm will receive the investigational drug NI-1801 at the P2RD every two weeks in combination with weekly administration of paclitaxel (80 mg/m^2) over 4-week cycles. The control arm will be treated with weekly paclitaxel at the same regimen.
  Arms: Randomized cohort
Drug: Paclitaxel — The control arm will be treated with weekly administration of paclitaxel (80 mg/m^2) over 4-week cycles.
  Arms: Randomized cohort

SUMMARY:
Study LCB-1801-001 is an open-label, Phase 1, dose escalation (Part A) and expansion (Part B), first-in-human clinical study of NI-1801 in patients with advanced, metastatic, or recurrent solid malignancies expressing mesothelin (MSLN).

The dose escalation part (Part A) of the main study will evaluate the safety and tolerability of escalating doses of NI-1801 to determine the maximum tolerated dose (MTD) and non-tolerated toxic dose (NTD) of NI-1801. The expansion part (Part B) of the main study will further evaluate the safety and efficacy of NI-1801 administered at or below the MTD in up to 10 additional subjects in order to determine the recommended Phase 2 dose (RP2D).

Treatments will be administered in 28-day cycles for up to 12 months until disease progression, unacceptable toxicity, or Investigator/patient decision to withdraw study consent.

The dose escalation part (Part A) of the sub-study will evaluate the safety and tolerability of escalating doses of NI-1801 in combination with anti-PD-1 antibody. The expansion part (Part B) of the sub-study will further evaluate the safety and efficacy of NI-1801 administered in combination with anti-PD-1 antibody at or below the MTD.

In the randomized cohort, the experimental arm will receive the investigational drug NI-1801 at the P2RD every two weeks in combination with weekly administration of paclitaxel (80 mg/m^2) over 4-week cycles. The control arm will be treated with weekly paclitaxel at the same regimen representing one of the standards of care (SoC) in this population. This trial specifically targets patients with platinum-resistant ovarian cancer. This cohort will be made up of 20 evaluable patients, 10 per arm.

ELIGIBILITY:
Main Inclusion Criteria for the Single Agent Dose Escalation and the Combination with Pembrolizumab:

1. Adults ≥ 18 years of age at the time of signing the informed consent form
2. Histologically or cytologically confirmed diagnosis of epithelial OC (high-grade serous or endometroid), TNBC, or non-squamous NSCLC. For the combination with pembrolizumab, only subjects with histologically or cytologically confirmed diagnosis of epithelial OC (high-grade serous or endometroid), non-squamous NSCLC and ductal pancreatic adenocarcinoma.
3. MSLN expression with staining intensity of ≥ 2+ as per IHC in ≥ 40% of tumor cells. Staining for MSLN expression can be performed using archival tumor tissue and is foreseen to be performed at the institution's pathology. A slice for centralized IHC assessment for validation and biomarker analysis is mandatory.
4. Patients with advanced, metastatic, or recurrent disease

   * after at least 1 prior systemic treatment for the primary malignancy and
   * who have failed treatment with, are intolerant to, or are not candidates for available therapies that are known to confer a clinical benefit to patients with these tumor entities.
5. Measurable disease according to the revised RECIST guideline version 1.1(3)
6. Patients treated in either the single agent recommended dose expansion cohort or in the combination with pembrolizumab cohort should have accessible lesions at screening for baseline and on treatment biopsies.
7. Eastern Cooperative Oncology Group performance status (ECOG PS) 0-1.
8. Negative pregnancy test at inclusion.
9. Life expectancy of at least 2 months.

Main Inclusion Criteria for the Randomized study arm:

1. Female patients ≥ 18 years of age.
2. Patients must have a confirmed diagnosis of high-grade serous epithelial ovarian cancer.
3. Patients must have platinum-resistant disease:

   3.1. Patients who have only had 1 line of platinum-based therapy must have received at least 4 cycles of platinum, must have had a response (CR or PR) and then progressed between greater than 3 months and ≤ 6 months after the date of the last dose of platinum.

   3.2. Patients who have received 2 or 3 lines of platinum therapy must have progressed on or within 6 months after the date of the last dose of platinum
4. Patients must have progressed radiographically on or after their most recent line of therapy.
5. Patients must be willing to provide an archival tumor tissue block or slides, or undergo procedure to obtain a new biopsy using a low risk, medically routine procedure for IHC confirmation of MSLN expression.
6. MSLN expression with staining intensity of ≥ 2+ as per IHC in ≥ 40% of tumor cells. Staining for MSLN expression can be performed using archival tumor tissue and can be done at the institution's pathology. A slice for centralized IHC assessment for validation and biomarker analysis is mandatory.
7. Patients must have at least one lesion that meets the definition of measurable disease by RECIST v1.1 (radiologically measured by the Investigator).
8. Patients must have received at least 1 but no more than 3 prior systemic lines of anticancer therapy, and for whom single-agent therapy is appropriate as the next line of treatment:

   * Adjuvant ± neoadjuvant considered one line of therapy
   * Maintenance therapy (e.g., bevacizumab, PARP inhibitors) will be considered as part of the preceding line of therapy (i.e., not counted independently)
   * Therapy changed due to toxicity in the absence of progression will be considered as part of the same line (i.e., not counted independently)
   * Hormonal therapy will be counted as a separate line of therapy unless it was given as maintenance
9. ECOG PS of 0 or 1
10. Time from prior therapy:

    * Systemic antineoplastic therapy (5 half-lives or 4 weeks, whichever is shorter)
    * Focal radiation completed at least 2 weeks prior to first dose of study drug
11. Patients must have stabilized or recovered (Grade 1 or baseline) from all prior therapy-related toxicities.
12. Major surgery must be completed at least 4 weeks prior to first dose and have recovered or stabilized from the side effects of prior surgery.
13. Patients must have adequate hematologic, liver and kidney functions
14. Patients or their legally authorized representative must be willing and able to sign the informed consent form (ICF) and to adhere to the protocol requirements.
15. Negative pregnancy test at inclusion

Main Exclusion Criteria for the Single Agent Dose Escalation and the Combination with Pembrolizumab:

1. Patient has known hypersensitivity to NI-1801 or any of the constituent compounds.
2. Radiotherapy to the target lesions within 4 weeks prior to the first NI-1801 infusion.
3. Prior anti-cancer therapy including chemotherapy, hormonal therapy, and investigational agents within 2 weeks or within ≤ 5 half-lives prior to starting NI-1801 dosing (up to a maximum of 4 weeks), whichever is longer. The maximum required washout period will thus not exceed 4 weeks prior to the day of first treatment with NI-1801. Note: Low dose steroids (oral prednisone or equivalent ≤ 20 mg per day, including systemic or topic use), localized noncentral nervous system (CNS) radiotherapy of non-target lesions, and treatment with bisphosphonates and RANKL inhibitors are not criteria for exclusion.
4. Other investigational therapies must not be used, i.e., treatment within another clinical trial is not permitted, while the patient is on study. COVID-19 vaccination is allowed only starting from Cycle 2 (if not completed before study inclusion).
5. Severe cardiac dysfunction (NYHA classification III-IV).
6. Significant hepatic dysfunction (serum bilirubin ≥ 1.5 mg/dL or AST and/or ALT ≥ 2.5 times normal level), unless related to liver metastasis.
7. Patients with known human immunodeficiency virus (HIV) infection or known history or serological evidence of prior hepatitis B or C virus infection. Active SARS-COV2 infection.
8. Uncontrolled active systemic bacterial, viral, fungal, or other infection (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment), or intravenous anti-infective treatment within 2 weeks prior to first dose of NI-1801.
9. Patients with concomitant active malignancy, requiring ongoing systemic treatment.
10. Patients with known CNS metastases.
11. Platelet count lower than 100 x 10^9/L (transfusion support within 14 days before the test is not allowed).
12. Hemoglobin lower than 10.0 g/dL. Prior RBC transfusion is permitted.
13. ANC lower than 1 x 10^9/L (the use of colony stimulating factors, G-CSF or GM-CSF, within 14 days before the test is not allowed).
14. Pregnancy and lactation.
15. History of psychiatric illness or substance abuse likely to interfere with ability to comply with protocol requirements or give informed consent.
16. Significant medical diseases or conditions, including laboratory abnormalities, as assessed by the Investigators and Sponsor, which would substantially increase the risk-benefit ratio of participating in the study. This includes, but is not limited to, acute myocardial infarction within the last 6 months, unstable angina, uncontrolled diabetes mellitus, and severely immunocompromised state, major surgery ≤ 4 weeks prior to starting NI-1801.
17. Prior treatment with a CD47, SIRPα, or MSLN targeting agent.
18. Patients in whom acute toxic effects of any prior radiotherapy, chemotherapy, or surgical procedure have not resolved to Grade ≤ 1 or returned to baseline except for alopecia (any grade), anemia, and peripheral neuropathy (for the latter, recovery to Grade ≤ 2 is acceptable).
19. People who are detained through a court or administrative decision, receiving psychiatric care against their will, adults who are the subject of a legal protection order (under tutorship/curatorship), people who are unable to express their consent, and people who are subject to a legal guardianship order.

Furthermore, subjects presenting with any of the following criteria will not be included in the sub-study (combination with pembrolizumab cohort):

* History of/active non-infectious pneumonitis or interstitial lung disease.
* Known hypersensitivity to pembrolizumab or excipients.
* Participants with an active, known or suspected autoimmune disease. Participants with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
* Prior organ or tissue allograft.
* History of Grade ≥ 3 toxicity related to prior T-cell agonist or checkpoint inhibitor therapy, except those that are unlikely to re-occur with standard countermeasures.
* History of myocarditis, regardless of etiology.

Main Exclusion Criteria for the Randomized study arm:

1. Patients with clear cell, mucinous, or sarcomatous histology, mixed tumors containing any of the above histology, or low-grade or borderline ovarian tumor.
2. Patients with primary platinum-refractory disease, defined as disease that did not respond to (CR or PR) or has progressed within 3 months of the last dose of first line platinum-containing chemotherapy.
3. Patients with prior wide-field radiotherapy (RT) affecting at least 20% of the bone marrow.
4. Patients with serious concurrent illness or clinically relevant active infection, including, but not limited to the following:

   * Active hepatitis B or C infection (whether or not on active antiviral therapy)
   * HIV infection
   * Active cytomegalovirus infection
   * Any other concurrent infectious disease requiring IV antibiotics within 2 weeks before starting study drug Note: Testing at screening is not required for the above infections unless clinically indicated
   * Patients with history of multiple sclerosis or other demyelinating disease and/or Lambert-Eaton syndrome (paraneoplastic syndrome)
5. Patients with clinically significant cardiac disease including, but not limited to, any one of the following:

   * Myocardial infarction ≤ 6 months prior to first dose
   * Unstable angina pectoris
   * Uncontrolled congestive heart failure (New York Heart Association greater than class II)
   * Uncontrolled ≥ Grade 3 hypertension (per CTCAE)
   * Uncontrolled cardiac arrhythmias
   * Patients assigned to PLD stratum only: Left ventricular ejection fraction (LVEF) below the institutional limit of normal as measured by echocardiography (ECHO) or multigated acquisition (MUGA) scan
   * History of hemorrhagic or ischemic stroke within six months prior to randomization
6. History of cirrhotic liver disease (Child-Pugh Class B or C)
7. Previous clinical diagnosis of non-infectious interstitial lung disease (ILD), including noninfectious pneumonitis
8. Patients with prior hypersensitivity to monoclonal antibodies.
9. Women who are pregnant or lactating.
10. Patients with prior treatment with a CD47, signal regulatory protein (SIRP) alpha, or MSLN targeting agent.
11. Patients with central nervous system (CNS) metastases.
12. Patients with a history of other malignancy within 3 years prior to randomization.
13. Prior known hypersensitivity reactions to study drugs and/or any of their excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-04-29 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT) | Up to 12 months
  Is defined as any of the toxicities occurring within the DLT window (Cycle 1, Days 1 to 28) except those that are clearly and incontrovertibly due to extraneous causes.
Non-Tolerated Dose (NTD) | Up to 12 months
  Is defined as a dose level at which 2 or more of up to 6 evaluable patients in a cohort experience a DLT in the 4-week DLT window.
Maximum Tolerated Dose (MTD) | Up to 12 months
  Is defined as the last cohort below the NTD with 0 or 1 out of 6 evaluable subjects experiencing a DLT during the 4-week DLT window.
Progression Free Survival (PFS) (Randomized Cohort only) | Up to 12 months
  Defined as the time from date of randomization until Investigator-assessed progressive disease or death, whichever occurs first.
Adverse Events (AEs) | Up to 12 months
  Number of patients with AEs as assessed by CTCAE v5.0

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Up to 12 months
  Is defined as the proportion of patients who achieve a partial response (PR) or better better, i.e., PR + complete response (CR), of the defined target lesions compared to baseline.
Disease Control Rate (DCR) | Up to 12 months
  Is defined as the proportion of patients who achieve a clinical benefit from NI-1801 treatment, i.e., CR + PR + stable disease (SD).
Best Overall Response (BOR) | Up to 12 months
  Is defined as the best response recorded from start of NI-1801 treatment until the first date that recurrent or progressive disease is objectively documented.
Time to Response | Up to 12 months
  Is defined as the time from the first NI-1801 dose date to the date of first documented response (i.e., PR or better)
Duration of Response | Up to 12 months
  Is defined as the time from the earliest date of documented response (i.e., CR or PR) to the first date that disease progression, recurrence of disease, or death, whichever occurs first, is objectively documented
Progression Free Survival | Up to 12 months
  Is defined as the time from the first dose of NI-1801 to progressive disease or death from any cause, whichever occurs first
Overall Survival | Up to 12 months
  Is defined as the time from the first dose of NI-1801 to death from any cause
Pharmacokinetics - Cmax | Up to 12 months
  Maximum concentration of drug
Pharmacokinetics - tmax | Up to 12 months
  Time to maximum concentration
Pharmacokinetics - t1/2 | Up to 12 months
  Terminal Half-life
Pharmacokinetics - AUC | Up to 12 months
  Area under the curve
Pharmacokinetics - CL | Up to 12 months
  Total body clearance
Presence of anti-drug antibodies (ADA) | Up to 12 months
  Detection of ADAs in patients
Frequency of anti-drug antibodies (ADA) | Up to 12 months
  Frequency of ADAs in patients
Functional impact of anti-drug antibodies (ADA) | Up to 12 months
  ADAs impact on Cmax and AUC as well as response variables
Biomarker CA125 (Randomized cohort only) | Up to 12 months
  Evaluate changes of CA125 levels compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, MD, Study Director — LCB - Novimmune SA
Locations (7):
- France (4):
  - Institut Curie, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - Centre Eugène Marquis, Rennes
  - Gustave Roussy, Villejuif, France
- Italy (3):
  - Humanitas Research Hospital, Milan
  - Istituto Europeo di Oncologia, Milan
  - Centro Ricerche Cliniche Verona, Verona

IPD SHARING:
Plan to Share IPD: No